CLINICAL TRIAL: NCT04792138
Title: Learning MRI and Histology Image Mappings for Cancer Diagnosis and Prognosis
Acronym: Histo-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 251440
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer; Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prostatectomy and biopsy specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men suspected of Prostate Cancer
  Interventions: Diagnostic Test: VERDICT MRI; Diagnostic Test: Luminal Index Imaging

INTERVENTIONS:
Diagnostic Test: VERDICT MRI — Advanced Diffusion Model
Diagnostic Test: Luminal Index Imaging — Advanced T2 mapping

SUMMARY:
Multiparametric magnetic resonance imaging (mpMRI) is now widely used to risk stratify men with a suspicion of prostate cancer and identify suspicious regions for biopsy. Advanced MRI techniques have emerged which seek to improve this characterisation and could predict biopsy results non-invasively before men undergo biopsy. Before these techniques are translated clinically, robust histological and clinical validation is required.

This study aims to clinically validate advanced MRI techniques in a cohort of men suspected with prostate cancer. Histological analysis of men undergoing biopsy, +/- prostatectomy will be used for biological validation of VERDICT; Vascular and Extracellular Restricted Diffusion for Cytometry in Tumours and Luminal Water imaging (LWI). In particular, prostatectomy specimens will be processed using 3-D printed patient-specific moulds to allow for accurate MRI and histology mapping.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-90 with a clinical suspicion of prostate cancer
* No contraindication to MRI

Exclusion Criteria

* Men unable to have a MRI scan, or in whom artefact would reduce quality of MRI
* Men unable to given informed consent
* Previous treatment (prostatectomy, radiotherapy, brachytherapy) of prostate cancer
* Ongoing hormonal treatment for prostate cancer

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity. Men with clinical suspicion of prostate cancer.
Study Population: Cohort of men presenting to our recruitment centre with suspicion of prostate cancer due to raised prostate specific antigen level or suspicious clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of VERDICT MRI | 2 years
  Quantitative assessment of VERDICT MRI reduces false positives by 10% compared to standard MRI alone
Diagnostic accuracy of Luminal Water Imaging (LWI) | 2 years
  Quantitative assessment of LWI reduces false positives by 10% compared to standard MRI alone

SECONDARY OUTCOMES:
The proportions of true positives with index tests is the same as mpMRI. | 2 years

OTHER OUTCOMES:
Machine learning algorithms can predict histology from MRI. | 3 years
  Number of correct predictions of gleason grade in men who undergo biopsy or prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Shonit Punwani, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh S, Mathew M, Mertzanidou T, Suman S, Clemente J, Retter A, Papoutsaki MV, Smith L, Grussu F, Kasivisvanathan V, Grey A, Dinneen E, Shaw G, Carter M, Patel D, Moore CM, Atkinson D, Panagiotaki E, Haider A, Freeman A, Alexander D, Punwani S. Histo-MRI map study protocol: a prospective cohort study mapping MRI to histology for biomarker validation and prediction of prostate cancer. BMJ Open. 2022 Apr 8;12(4):e059847. doi: 10.1136/bmjopen-2021-059847. PMID 35396316